CLINICAL TRIAL: NCT04964154
Title: Building Resiliency and Vital Equity (BRAVE) Project: Understanding Native Americans' Perceptions/Beliefs About COVID-19 Testing and Vaccination Study
Acronym: BRAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Carolina Central University (Other)
Collaborators: Lumbee Tribe of North Carolina (Unknown); University of North Carolina at Pembroke (Unknown)
Responsible Party: Principal Investigator, Deepak Kumar, Director of Julius L. Chambers Biomedical/Biotechnology Research Institute, North Carolina Central University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1201571
Record Dates: First submitted 2021-07-13; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Covid19 Virus Infection
Keywords: COVID-19 testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive information about testing and vaccination based on zip code.
Masking Description: No masking employed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRAVE Non-Intervention (No Intervention): Survey participants in the BRAVE non-intervention arm will not have received information (e.g., informational pamplets, flyers, townhalls) about COVID-19 testing and vaccination from the BRAVE project.
- BRAVE Intervention (Active Comparator): Survey participants in the BRAVE intervention arm will have received information (e.g., informational pamplets, flyers, townhalls) about COVID-19 testing and vaccination from the BRAVE project.
  Interventions: Behavioral: Protect Your Elders Campaign

INTERVENTIONS:
Behavioral: Protect Your Elders Campaign — This is a behavioral intervention where participants will receive cultural appropriate educational information about COVID-19 testing and vaccination.
  Arms: BRAVE Intervention

SUMMARY:
The Building Resilience and Vital Equity (BRAVE) project seeks to partner with American Indian tribal communities in North Carolina to establish COVID-19 services and resources for American Indian communities. The goal of this study is to 1) understand the barriers and social implications of COVID19 testing and vaccination among American Indians by designing and implementing culturally sensitive survey tools and intervention materials; 2) Implement BRAVE outreach and testing interventions to increase testing in American Indian communities; 3) analyze data and share back with tribal communities to improve perceptions of COVID-19 testing in the AI community and decrease in vaccine hesitancy.

ELIGIBILITY:
Inclusion Criteria:

- Self reports as Native American or American Indian

Exclusion Criteria:

* Does not self-report as Native American or American Indian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase in COVID-19 testing | 1 month
  Survey responses to determine if participants in zipcodes selected for intervention are more less inclined to get tested for COVID-19.
Increase in COVID-19 vaccination | 1 month
  Survey responses to determine if participants in zipcodes selected for intervention are more less inclined to get vaccinated against COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kumar, PhD, Principal Investigator — North Carolina Central University
Locations (1):
- Lumbee Tribe Tribal Housing Complex, Pembroke, North Carolina, United States